CLINICAL TRIAL: NCT05100225
Title: A Multiple Arm, Multicenter, Prospective, Randomized, Double-Blind, Placebo-Controlled, Parallel-Arm, Phase 2 Study of Intra-Articular Administration of an Allogeneic Human Placental Tissue Particulate (PTP-001) for the Treatment of Knee Osteoarthritis
Brief Title: Efficacy and Safety Trial of PTP-001 (MOTYS) for Symptomatic Knee Osteoarthritis
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Bioventus LLC (Industry)
Collaborators: NBCD A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KOA-21-02
Record Dates: First submitted 2021-10-19; First posted 2021-10-29 (Actual); Last update posted 2022-07-19 (Actual); Status verified 2022-07

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: A Multiple Arm, Multicenter, Prospective, Randomized, Double-Blind, Placebo-Controlled, Parallel-Arm, Phase 2 Study
Who Masked: Participant, Investigator
Masking Description: This is a double-blinded trial, in which neither participant nor investigator will know the content of the investigational product. Additionally, the study staff preparing the syringe. The unblinded personnel must not be involved in any other operational aspects of the trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- PTP-001 200 mg (Experimental): A single intra-articular injection in the target knee of PTP-001 200 mg.
  Interventions: Biological: PTP-001
- PTP-001 100 mg (Experimental): A single intra-articular injection in the target knee of PTP-001 100 mg.
  Interventions: Biological: PTP-001
- Placebo/saline (Placebo Comparator): A single intra-articular injection in the target knee of 4mL of placebo control - physiological saline (0.9% sodium chloride injection, USP).
  Interventions: Other: Placebo control

INTERVENTIONS:
Biological: PTP-001 — Allogeneic human placental tissue particulate (PTP-001) is administered as a single intra-articular injection to the target knee after resuspension with saline.
  Arms: PTP-001 100 mg; PTP-001 200 mg
Other: Placebo control — The placebo control, physiological saline (0.9% sodium chloride injection, USP), is administered as an intra-articular injection to the target knee.
  Other Names: Physiological saline
  Arms: Placebo/saline

SUMMARY:
Evaluation of safety, tolerability and efficacy of a single intra-articular (IA) injection of PTP-001, an allogeneic placental tissue particulate, in individuals with knee osteoarthritis (OA).

DETAILED DESCRIPTION:
This is a multiple arm, multicenter, prospective, randomized, double-blind, placebo-controlled, parallel-arm, phase 2 study of intra-articular administration of an allogeneic human placental tissue particulate (PTP-001) for the treatment of knee osteoarthritis. The study is planned to be conducted outside the United States. A total of approximately 210 participants are planned to be randomized to receive 1 of 2 doses of PTP-001 (100 mg or 200 mg) or saline vehicle control (placebo) injection. The purpose of the trial is to evaluate the efficacy, safety and tolerability of a single low dose and high dose of PTP-001 compared to placebo over a 26-week period.

ELIGIBILITY:
Inclusion Criteria:

* Participants are eligible to be included in the study only if all of the following criteria apply:

  1. Male or female, aged 40 to 80 years
  2. Symptomatic knee OA with Kellgren-Lawrence radiographic classification of 2 or 3 (mild or moderate) as assessed by the central reading facility
  3. Target knee pain ≥ 20 and ≤ 40 out of 50 the WOMAC®NRS 3.1 pain questionnaire (sum of 5 questions) at screening and baseline
  4. Onset of symptomatic OA of the target knee was at least 6 months prior to screening
  5. Insufficient or failed response or intolerance to analgesics and/or non-steroidal anti-inflammatory drugs, as reported by the participant
  6. IF FEMALE, must meet all of the following:

     * Not breast feeding
     * Not planning to become pregnant during the study
     * If of childbearing potential, must have a negative pregnancy test result within 72 hours prior to receiving the intra-articular injection, and must commit to the use of a highly effective form of birth control (See Appendix A) for at least 12 weeks after the injection
  7. Willingness to remain on the same oral "rescue" (as needed) analgesic as the only pharmacologic treatment for knee pain during the study
  8. Willingness to abstain from taking any illicit or unauthorized medications for treatment of OA or any other concurrent condition during the study
  9. Written informed consent is obtained from the participant

Exclusion Criteria:

* Participants are excluded from the study if any of the following criteria apply:

  1. Participant is non-ambulatory (unable to walk >50 feet without assistance)
  2. Clinically severe obesity as defined by the National Institutes of Health (body mass target ≥40 kg/m2)
  3. Contralateral knee pain equal to or exceeding the pain in the target knee (on the WOMAC® NRS3.1 pain questionnaire) at screening and/or baseline
  4. Clinically significant effusion of the target knee at either the screening or baseline visits determined by physical examination (e.g., ballotable patella or positive bulge sign). Note: Participants presenting with effusion may be enrolled in the study after undergoing knee aspiration to remove excess fluid in the target joint.
  5. Severe (excessive) malalignment of the tibial-femoral axis, assessed radiographically
  6. Presence of active infection of the target knee or systemic infection requiring treatment within the 3 months prior to screening
  7. Clinical diagnosis of inflammatory arthritis (e.g., rheumatoid arthritis, psoriatic arthritis, ankylosing spondylitis, systemic lupus erythematosus, etc.) established by clinical history, examination, or serology
  8. Participant is receiving, has received, or plans to receive any of the following therapies

     * Prior administration of hyaluronic acid, extended release corticosteroid (e.g., Zilretta®), platelet-rich plasma (PRP), or stem cell therapies by intra-articular injection(s) of the target knee within 6 months prior to screening
     * Prior intra-articular corticosteroid within 3 months prior to screening or into any other joint within 30 days prior to screening
     * Current chronic systemic use of corticosteroids in doses exceeding 10 mg prednisolone-equivalents daily
     * Treatment with any investigational therapy (drug, device, or biologic) within 3 months prior to screening or is planned for the duration of the study
     * Treatment with immunosuppressive medication or chemotherapy within the past 5 years
  9. Chronic use of narcotics or alcohol abuse within the past 6 months prior to screening
  10. Surgery to the target knee (including arthroscopy) within 6 months prior to receiving the intra-articular injection or planned surgery to the target knee within 6 months after the injection
  11. Participant previously underwent arthroplasty of the target knee
  12. Presence of joint instability or complaints of locking, intermittent limitation in range of motion, or loose body sensation, suggestive of internal derangement of the knee (either extremity)
  13. Symptomatic OA of the non-target knee that is not responsive to paracetamol (acetaminophen) or oral nonsteroidal anti-inflammatory drugs (NSAIDs).
  14. Diagnosis of lower extremity gout or pseudo-gout in the past 6 months
  15. Osteonecrosis of either knee
  16. Significant acute (within the past 3 months) injury to the target knee
  17. History of receiving a solid organ or hematologic transplant
  18. History of malignancy, radiotherapy, or chemotherapy for malignancy within the past 5 years, except for basal or squamous cell carcinoma of the skin
  19. History of prior radiation therapy of the target knee
  20. History of autoimmune disease affecting the musculoskeletal system
  21. Known (documented) history of acquired immune deficiency syndrome or human immunodeficiency virus
  22. Any condition causing pain in or around the target knee (e.g., radiating pain, pain in another region of the ipsilateral lower extremity) that may interfere with assessment(s) of the target knee
  23. Other chronic pain anywhere in the body that requires the chronic use of analgesic medications, such as fibromyalgia, neuropathic pain, low back pain, etc.
  24. Presence of contraindications for use of 3 g/day of orally administered paracetamol/acetaminophen due to known hypersensitivity or hepatic impairment.
  25. Known presence of any concurrent medical condition (e.g., hematologic renal, hepatic, cardiac, or coagulation abnormalities) that in the investigator's judgment would interfere with the required study assessments and study participation
  26. Participant is involved in litigation (e.g., worker's compensation) for a medical condition or injury at any anatomical site

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2021-09-30 (Actual); Primary Completion 2022-10-31 (Estimated); Study Completion 2022-11-30 (Estimated)

PRIMARY OUTCOMES:
Efficacy - Change from pretreatment baseline in the WOMAC pain subscale | At 6 months
  To evaluate the change from pretreatment baseline in the WOMAC pain sub-score in the target knee on an 11-box numerical rating scale, with categories from 0 (none) to 10 (extreme), normalized on scales of 0-100.
Safety - Incidence of local and systemic AEs | Over 6 months
  To assess the long-term (6 months) incidence of local and systemic AEs, and consists of physical examination, laboratory values, AEs, AESI, and immunogenicity testing.

SECONDARY OUTCOMES:
Change from pretreatment baseline in pain intensity assessed by participant self report (WOMAC Pain subscale). | At 2 weeks, 3 months, 4 months, 5 months.
  WOMAC Numerical Rating Scale (NRS) 3.1 questionnaire is a health status measure questionnaire of 24 questions comprising 3 subscales (pain, stiffness and physical function). WOMAC A (measure of pain) is measured on an 11-box numerical rating scale, with categories from 0 (none) to 10 (extreme), normalized to a scale of 0-100, where higher score represents higher pain.
Change from pretreatment baseline in function assessed by participant self-report (WOMAC Function subscale). | At 2 weeks, 3 months, 4 months, 5 months, and 6 months.
  WOMAC Numerical Rating Scale (NRS) 3.1 questionnaire is a health status measure questionnaire of 24 questions comprising 3 subscales (pain, stiffness and physical function). WOMAC C (measure of physical function) is measured on 11-point NRS ranging from 0 (none) to 10 (extreme), where higher score represents higher difficulties in physical function.
Change from pretreatment baseline in the weekly average of daily pain assessed by patient self report (NRS). | At 2 weeks, 3 months, 4 months, 5 months, and 6 months.
  The question is an average daily (24-h) pain intensity score on a 0 to 10 NRS scale with 0 indicating 'no pain' and 10 indicating 'pain as bad as you can imagine'.
Change from pretreatment baseline in patient global assessment of OA (PGA-OA) assessed by participant self report. | At 2 weeks, 3 months, 4 months, 5 months, and 6 months.
  Considering all the ways knee osteoarthritis affects the participants, the question is an average daily (24-h) self-reported global assessment on an 11-box numerical rating scale, with 0 indicating "very good" and 10 indicating "very poor".
Change from pretreatment baseline in participant self-reported quality of life measured by SF-36 overall score, PCS, and MCS. | At 3 months and 6 months.
  The SF-36 measures 8 domains: physical functioning, role physical, bodily pain, general health, vitality, social functioning, role emotional, and mental health, and has 2 summary scores (physical and mental). The physical health measure includes 4 scales of physical functioning (10 items), role-physical (4 items), bodily pain (2 items), and general health (5 items). The mental health measure is composed of vitality (4 items), social functioning (2 items), role-emotional (3 items), and mental health (5 items).
  The assessment is performed on a scale of 0 (maximum disability)-100 (no disability) with higher scores indicating better health status.
Response to PTP-001 on the OMERACT-OARSI responder criteria. | At 2 weeks, 3 months, and 6 months.
  The OMERACT-OARSI responder criteria involve changes that are deemed to be clinically relevant in the three domains: pain, function, and Patient Global Assessment. For each of these domains, ranges are defined for absolute and percent changes from baseline that correspond to "high improvement" and "moderate improvement". OMERACT-OARSI response is defined as either i) improvement in pain or physical function ≥50% and an absolute change ≥20 mm on a 100-mm visual analog scale; or (2) improvement of ≥20% and with an absolute change ≥10 mm in at least two of the following three categories: pain, physical function, and patient's global assessment (PGA).

CONTACTS AND LOCATIONS:
Overall Officials: Moin Khan, MD, Principal Investigator — McMaster University Department of Surgery St. Joseph's Healthcare Hamilton
Locations (14):
- Australia (5):
  - Emeritus Research Sydney, Botany, New South Wales
  - Genesis Research Services, Broadmeadow, New South Wales
  - Royal North Shore Hospital, Saint Leonards, New South Wales
  - Holdsworth House Medical Practice, Sydney, New South Wales
  - Emeritus Research Melbourne, Camberwell, Victoria
- Canada (6):
  - Hamilton Medical Research Group, Hamilton, Ontario
  - McMaster University Department of Surgery St. Joseph's Healthcare Hamilton, Hamilton, Ontario
  - Canadian Phase Onward Inc., Toronto, Ontario
  - Diex Recherche Quebec Inc., Québec, Quebec
  - Centrede Recherche Saint-Louis, Québec, Quebec
  - Diex Recherche Sherbrooke Inc., Sherbrooke, Quebec
- Denmark (3):
  - Sanos Clinic Nordjylland, Gandrup
  - Sanos Clinic, Herlev
  - Sanos Clinic Syddanmark, Vejle

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Flannery CR, Seaman SA, Buddin KE, Nasert MA, Semler EJ, Kelley KL, Long M, Favret J, Pavesio A, Loeser RF. A novel placental tissue biologic, PTP-001, inhibits inflammatory and catabolic responses in vitro and prevents pain and cartilage degeneration in a rat model of osteoarthritis. Osteoarthritis Cartilage. 2021 Aug;29(8):1203-1212. doi: 10.1016/j.joca.2021.03.022. Epub 2021 May 20. PMID 34023528